CLINICAL TRIAL: NCT05548972
Title: Global, Multicenter and Prospective Post-Market Clinical Follow-Up Study of the G7® Dual Mobility Acetabular System With Vivacit-E® or Longevity® Poly Bearing & Instrumentation
Brief Title: G7 Dual Mobility With Vivacit-E or Longevity PMCF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMG2020-42H
Record Dates: First submitted 2022-09-07; First posted 2022-09-22 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Hip Osteoarthritis; Rheumatoid Arthritis; Joint Diseases; Avascular Necrosis; Dislocation, Hip; Femoral Neck Fractures; Trochanteric Fractures; Revision Surgeries
Keywords: Total Hip arthroplasty; Revision Hip arthroplasty; Medical device; Safety; Performance; Clinical benefit; G7 Dual Mobility
MeSH Terms: conditions — Osteoarthritis, Hip; Arthritis, Rheumatoid; Joint Diseases; Osteonecrosis; Hip Dislocation; Femoral Neck Fractures; Hip Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- G7 Dual Mobility with Vivacit-E polyethylene bearing in primary THA (Other): Subjects in need of a total hip arthroplasty who meet inclusion/exclusion criteria (anticipated enrollment: 60)
  Interventions: Device: G7 Dual Mobility with Vivacit-E bearing
- G7 Dual Mobility with Vivacit-E polyethylene bearing in revision (total) hip arthroplasty (Other): Subjects in need of a revision (total) hip arthroplasty who meet inclusion/exclusion criteria (anticipated enrollment: 119)
  Interventions: Device: G7 Dual Mobility with Vivacit-E bearing
- G7 Dual Mobility with Longevity polyethylene bearing in primary THA (Other): Subjects in need of a total hip arthroplasty who meet inclusion/exclusion criteria(anticipated enrollment: 60)
  Interventions: Device: G7 Dual Mobility Longevity bearing
- G7 Dual Mobility with Vivacit-E Longevity bearing in revision (total) hip arthroplasty (Other): Subjects in need of a revision (total) hip arthroplasty who meet inclusion/exclusion criteria (anticipated enrollment: 119)
  Interventions: Device: G7 Dual Mobility Longevity bearing

INTERVENTIONS:
Device: G7 Dual Mobility with Vivacit-E bearing — hip arthroplasty with G7 Dual Mobility Vivacit-E bearing
  Arms: G7 Dual Mobility with Vivacit-E polyethylene bearing in primary THA; G7 Dual Mobility with Vivacit-E polyethylene bearing in revision (total) hip arthroplasty
Device: G7 Dual Mobility Longevity bearing — hip arthroplasty with G7 Dual Mobility Longevity bearing
  Arms: G7 Dual Mobility with Longevity polyethylene bearing in primary THA; G7 Dual Mobility with Vivacit-E Longevity bearing in revision (total) hip arthroplasty

SUMMARY:
This study is a global, multi-center, prospective, non-controlled, non-randomized, post-market clinical follow-up study. The main objectives of this study are to confirm the long-term safety, performance, and clinical benefits of the G7 Dual Mobility Acetabular System when used with the Vivacit-E or Longevity polyethylene hip bearing and instrumentation in primary total and revision (total) hip arthroplasty

DETAILED DESCRIPTION:
The G7 Dual Mobility construct offers dislocation resistance without the need to constrain the femoral head, providing stability and high range of motion. Dual Mobility systems decrease the risk of post-operative instability in high-risk patients in both primary and revision arthroplasties.

This study will enroll up to 358 hips globally, 179 for the Vivacit-E and 179 for the Longevity polyethylene bearings. From the 179 hips per bearing variant, the study will enroll 60 primary and 119 revision arthroplasty hips. The Longevity bearing variant will only be enrolled in the US, as it is not CE marked and unregistered in the APAC market. Vivacit-E bearings will be enrolled globally.

A maximum of 20 study centers will be selected globally. To minimize potential bias and to maximize our ability to assess inter-site differences, each study site will target maximum 24 primary hip arthroplasties and maximum 47 revision hip arthroplasties. Each site is encouraged to enroll both, primary and revision, subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 to 80 years of age, inclusive
* Patient is skeletally mature
* Patient qualifies for (total) hip arthroplasty based on physical exam and medical history including at least one of the following:

  * Non-inflammatory degenerative joint disease, including osteoarthritis and avascular necrosis
  * Rheumatoid arthritis
  * Dislocation risks
  * Correction of functional deformity
  * Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques
  * Revision procedures where other treatment or devices have failed.
* Patient is willing and able to complete scheduled follow-up evaluations as described in the protocol and Informed Consent
* Patient, or the patient's legally authorized representative (LAR), has participated in the Informed Consent process and is willing and able to sign an IRB/EC approved Informed Consent

Exclusion Criteria:

* Patient is septic, has an active infection or has osteomyelitis at the affected joint
* Patient has significant osteoporosis as defined by treating surgeon
* Patient has metabolic disorder(s) which may impair bone formation
* Patient has osteomalacia
* Patient has distant foci of infections which may spread to the implant site
* Patient has rapid joint destruction, marked bone loss or bone resorption apparent on pre-operative radiographs
* Patient underwent contralateral THA within 3 months of planned index procedure or has a contralateral THA planned within 3 months of the index procedure
* Patient is undergoing simultaneous bilateral THA
* Patient has vascular insufficiency, muscular atrophy at the implant site or neuromuscular disease which are likely to jeopardize the outcome of the surgery.
* Patient has any concomitant disease which is likely to jeopardize the functioning or success of the implant
* Patient is known to be pregnant
* The patient is in a vulnerable population group such as:

  * a prisoner
  * a known alcohol or drug abuser
  * mentally incompetent or unable to understand what participation in this study entails

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2037-01 (Estimated); Study Completion 2037-08 (Estimated)

PRIMARY OUTCOMES:
Survival of the implant system | 10 years
  Survival of the implant system based on removal of the study device
Safety of the implant system | 10 years
  Safety of the system will be assessed by monitoring the frequency and incidence of adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.

SECONDARY OUTCOMES:
Modified Harris Hip Score | 10 years
  The modified Harris Hip Score measures pain, function and functional activities using a self assessment. The overall score runs from 0-100 with 100 representing the best outcome.
Oxford Hip Score | 10 years
  The Oxford Hip Score measures pain and function using a self assessment. The overall score runs from 0-48 with 48 representing the best outcome.
EQ-5D-5L | 10 years
  The EQ-5D-5L measures the quality of life using a self assessment. The questionnaire includes 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Radiographic Assessment | 5 years
  X-ray evaluation to find significant radiographic findings such as radiolucency, osteolysis, atrophy, hypertrophy, component migration, device fracture, heterotopic ossification, etc

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Achakri, Study Director — Zimmer Biomet
Locations (10):
- United States (6):
  - Bowen Hefley Orthopedics, Little Rock, Arkansas
  - HCA HealthONE Orthopedic Specialists, Denver, Colorado
  - Jersey City Medical Center, Jersey City, New Jersey
  - Hospital for Special Surgery, New York, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - Slocum Research & Education Foundation, Eugene, Oregon
- UZ Leuven, Leuven, Belgium
- Istituto San Siro, Milan, Italy
- South Korea (2):
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do

IPD SHARING:
Plan to Share IPD: No